CLINICAL TRIAL: NCT05598164
Title: Botulinum Toxin Type A in the Treatment of Chronic Anal Fissure Without Excision
Brief Title: Botulinum Toxin Type A in the Treatment of Chronic Anal Fissure
Acronym: BTATCAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56IG701SSCC979
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-09

CONDITIONS: Chronic Anal Fissure
Keywords: Fissure in Ano; Anal fissure; botulinum toxin A; Chronic anal pain; Fecal incontinence; Spasm of the internal sphincter; Anal sphincter insufficiency
MeSH Terms: conditions — Fissure in Ano; Fecal Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Parallel Assignment A comparative, randomized, prospective, single-center clinical study. Patients of the main group are treated with injection in internal sphincter Botulinum toxin type A.
  In the control group, the fissure is excised in combination with a injection in internal sphincter Botulinum toxin type A with excision.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- main group (Experimental): Patients of main group are treated with injection in internal sphincter Botulinum toxin type A.
  Interventions: Other: Botulinum toxin type A
- control group (Experimental): In the control group, the fissure is excised in combination with a injection in internal sphincter Botulinum toxin type A.
  Interventions: Other: Botulinum toxin type A

INTERVENTIONS:
Other: Botulinum toxin type A — Patients of main group are treated with injection in internal sphincter botulinum toxin type A.
  In the control group, the fissure is excised in combination with a injection in internal sphincter botulinum toxin type A.

SUMMARY:
This study is aimed at studying the effectiveness and safety of surgical treatment of chronic anal fissure.

DETAILED DESCRIPTION:
A chronic anal fissure is a rupture of the mucous membrane of the anal canal, lasting more than 2 months and resistant to non-surgical treatment. This condition is accompanied by a strong pain syndrome during and after defecation (defecation). This condition is most often found in young and able-bodied adults, so the issue of treatment is of particular relevance.

The main cause of the development of a chronic anal fissure is a spasm of the internal sphincter. It should be eliminated first of all to ensure effective therapy. All the main treatment methods, such as medicinal relaxation of the internal sphincter with 0.4% nitroglycerin ointment, lateral subcutaneous sphincterotomy, and pneumodivulsion of the anal sphincter are aimed at its removal. However, the optimal method has not yet been developed.

Non-surgical treatments are often attended by relapse of disease, while surgical treatment is often complicated by intestinal contents incontinence, usually gas and loose or hard stool in some occasions (grade 3 anal sphincter insufficiency).

In particular, lateral subcutaneous sphincterotomy performed in such patients is associated with an increase in the degree of anal incontinence in the early post-operative period.

Botulinum Toxin Type A application in treatment of patients with chronic anal fissure (after fissure excision) is intended to improve the therapy results, namely to reduce the frequency and duration of anal sphincter insufficiency after sphincter spasm removal (reduction in the number of patients suffering from post-operative incontinence).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic anal fissure with spasm of anal sphincter

Exclusion Criteria:

* Inflammatory diseases of the colon
* Pectenosis
* Previous surgical interventions on the anal canal
* IV grade internal and external hemorrhoids
* Rectal fistula
* Severe somatic diseases at the decompensation stage
* Pregnancy and lactation
* Anal sphincter insufficiency
* Chronic paraproctitis
* Fibrous polyp of the anal canal, accompanied by clinical manifestations
* Individual intolerance and hypersensitivity to botulinum toxin
* Myasthenia gravis and myasthenic syndromes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Anal sphincter insufficiency | Up to 60 days
  Frequency of anal sphincter insufficiency according to the Wexner scale

SECONDARY OUTCOMES:
2-item pain intensity (P2) | On day 7, 30 and 60
  Self reported pain intensity after the defecation and during the day after the surgical intervention. Each item is scored 0-10 (0 = no pain; 10 = pain as bad, as can can be).
Non-Healing Wound | On day 15, 30, 45, 60
  Frequency of post-operative wound epithelialization
Profilometry /sphincterometry findings | On day 30, 60 and 365
  Internal sphincter spasm or local internal sphincter spasm by the data of anorectal profilometry / or anorectal sphincterometry
Temporary disability | Up to 60 days
  Duration of temporary disability
Relap | Up to 60 days
  Frequency of relapses

CONTACTS AND LOCATIONS:
Overall Officials: Sergey A. Frolov, Ph.D., Principal Investigator — State Scientific Centre of Coloproctology, Russian Federation (SSCCRussia)
Locations (1):
- SSCCRussia, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jorge JM, Wexner SD. Anorectal manometry: techniques and clinical applications. South Med J. 1993 Aug;86(8):924-31. doi: 10.1097/00007611-199308000-00016. PMID 8351556
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Nelson RL, Thomas K, Morgan J, Jones A. Non surgical therapy for anal fissure. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD003431. doi: 10.1002/14651858.CD003431.pub3. PMID 22336789
- [Background] Zetterstrom J, Mellgren A, Jensen LL, Wong WD, Kim DG, Lowry AC, Madoff RD, Congilosi SM. Effect of delivery on anal sphincter morphology and function. Dis Colon Rectum. 1999 Oct;42(10):1253-60. doi: 10.1007/BF02234209. PMID 10528760
- [Background] Delechenaut P, Leroi AM, Weber J, Touchais JY, Czernichow P, Denis P. Relationship between clinical symptoms of anal incontinence and the results of anorectal manometry. Dis Colon Rectum. 1992 Sep;35(9):847-9. doi: 10.1007/BF02047871. PMID 1511644
- [Background] Chen HL, Woo XB, Wang HS, Lin YJ, Luo HX, Chen YH, Chen CQ, Peng JS. Botulinum toxin injection versus lateral internal sphincterotomy for chronic anal fissure: a meta-analysis of randomized control trials. Tech Coloproctol. 2014 Aug;18(8):693-8. doi: 10.1007/s10151-014-1121-4. Epub 2014 Feb 6. PMID 24500725
- [Background] Valizadeh N, Jalaly NY, Hassanzadeh M, Kamani F, Dadvar Z, Azizi S, Salehimarzijarani B. Botulinum toxin injection versus lateral internal sphincterotomy for the treatment of chronic anal fissure: randomized prospective controlled trial. Langenbecks Arch Surg. 2012 Oct;397(7):1093-8. doi: 10.1007/s00423-012-0948-2. Epub 2012 Mar 20. PMID 22430300
- [Background] Bobkiewicz A, Francuzik W, Krokowicz L, Studniarek A, Ledwosinski W, Paszkowski J, Drews M, Banasiewicz T. Botulinum Toxin Injection for Treatment of Chronic Anal Fissure: Is There Any Dose-Dependent Efficiency? A Meta-Analysis. World J Surg. 2016 Dec;40(12):3064-3072. doi: 10.1007/s00268-016-3693-9. PMID 27539490
- [Background] Gui D, Cassetta E, Anastasio G, Bentivoglio AR, Maria G, Albanese A. Botulinum toxin for chronic anal fissure. Lancet. 1994 Oct 22;344(8930):1127-8. doi: 10.1016/s0140-6736(94)90633-5. PMID 7934496
- [Background] Stewart DB Sr, Gaertner W, Glasgow S, Migaly J, Feingold D, Steele SR. Clinical Practice Guideline for the Management of Anal Fissures. Dis Colon Rectum. 2017 Jan;60(1):7-14. doi: 10.1097/DCR.0000000000000735. No abstract available. PMID 27926552